CLINICAL TRIAL: NCT04661943
Title: Maintenance Therapy of Chidamide in Patients With HBV Positive Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: oubai (Other)
Responsible Party: Sponsor-Investigator, oubai, M.D., The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDB0369
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): Chidamide Specification: 5mg / tablet. Dosage: oral, 20 mg (3 tablets) each time, twice a week, with the interval of no less than 3 days (such as Monday and Thursday, Tuesday, Friday, Wednesday and Saturday, etc.)
  Interventions: Drug: Tucidinostat

INTERVENTIONS:
Drug: Tucidinostat — Tucidinostat Specification: 5mg / tablet. Dosage: oral, 20 mg (3 tablets) each time, twice a week, with the interval of no less than 3 days (such as Monday and Thursday, Tuesday, Friday, Wednesday and Saturday, etc.)
  Other Names: Chidamide，CS055，HBI-8000

SUMMARY:
A phase II，single arm，open-label study to assess Maintenance Therapy of Chidamide in Patients With Hepatitis B Virus（HBV）Positive Diffuse Large B-cell Lymphoma with complete response after completion of prior chemotherapy

DETAILED DESCRIPTION:
Objective to evaluate the efficacy and safety of maintenance therapy with Chidamide in patients With Hepatitis B Virus（HBV）Positive Diffuse Large B-cell Lymphoma（DLBCL） with complete response after completion of prior chemotherapy, so as to provide the basis for the application of Chidamide in HBV positive DLBCL

ELIGIBILITY:
Inclusion Criteria:

* histopathology confirmed DLBCL，with chronic hepatitis B before treatment
* After systemic treatment, complete response has been achieved and complete response lasted within 1year before enrollment
* The expected chemotherapy was completed and the laboratory indexes returned to normal
* The absolute value of neutrophil ≥ 1.5 × 10 9 / L, platelet count≥ 90 × 10 9 / L, hemoglobin level≥ 90 g / L
* Patients who cannot undergo hematopoietic stem cell transplantation for various reasons
* 18-75 years old, both male and female
* ECOG PS 0-1
* Body weight: male 67 ± 20 kg (47-87 kg), female 55 ± 20 kg (35-75 kg)
* expected survival time ≥3 months
* Voluntary written informed consent prior to trail screening

Exclusion Criteria:

* Pregnant and lactating women and women of childbearing age who are unwilling to take contraceptive measures
* Patients with prolonged QTc interval (male > 450ms, female > 470ms), ventricular tachycardia (VT), atrial fibrillation (AF), heart block, myocardial infarction (MI) within 1 year, congestive heart failure (CHF), and coronary heart disease with symptoms requiring drug treatment
* B-ultrasound showed that the width of the fluid dark area in the pericardial cavity was ≥ 10 mm at the end of diastolic period
* Patients with previous or planned organ transplantation
* Patients receiving symptomatic treatment for early myelotoxicity within 7 days before enrollment
* HBV nucleic acid quantitation > 103 IU / ml
* Patients with active bleeding
* Patients with thrombosis, embolism, cerebral hemorrhage, cerebral infarction and other this kind of diseases or medical history
* Patients with active infection or persistent fever within 14 days before enrollment
* less than 6 weeks after major organ surgery
* Abnormal liver function [total bilirubin > 1.5 times of the upper limit of normal value; ALT / AST > 2.5 times of upper limit of normal value for patients without liver metastasis ; ALT / AST > 5 times of upper limit of normal value for patients with liver metastasis ], abnormal renal function (serum creatinine > 1.5 times of upper limit of normal value)
* Mental disorders/Those who cannot obtain informed consent
* Patients with drug abuse and long-term alcohol abuse that affect evaluation
* The investigator determined not suitable to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 6months
  Progression-free survival（by IWC）

SECONDARY OUTCOMES:
Overall survival | 12months
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No